

# **Non-Interventional Study Protocol**

Protocol No:X9001260

Retrospective analysis to characterize the real world use patterns, efficacy and safety of ceftazidime-avibactam in the management of gram negative infections.

Statistical Analysis Plan (SAP)

Version: Draft Version 1.0

Author: PPD

**Date**: 10-Nov-2021

## TABLE OF CONTENTS

| 1 | AM | ENDMENTS FROM PREVIOUS VERSION(S) | 3 |
|----|-------|-----------------------------------------------|----|
| 2 | INT | RODUCTION | 3 |
| | 2.1 | Study Design | 3 |
| | Stud | y population | |
| | | i source | |
| | | tment/cohort labels | |
| | 2.2 | STUDY OBJECTIVES | 4 |
| 3 | HYI | POTHESES AND DECISION RULES | 5 |
| | 3.1 | STATISTICAL HYPOTHESES | 5 |
| | 3.2 | STATISTICAL DECISION RULES | 5 |
| 4 | ANA | ALYSIS SETS/POPULATIONS | 5 |
| | 4.1 | ALL SUBJECTs SET | 5 |
| | 4.2 | SAFETY ANALYSIS SET | |
| | 4.3 | OTHER ANALYSIS SET | 5 |
| | 4.4 | SUBGROUPS | 5 |
| 5 | ENI | POINTS AND COVARIATES | 5 |
| | 5.1 | Efficacy/Effectiveness Endpoint(s) | 5 |
| | 5.2 | SAFETY ENDPOINTS | |
| | 5.3 | OTHER ENDPOINTS | 6 |
| | 5.4 | Covariates | 6 |
| 6 | HAN | NDLING OF MISSING VALUES | 6 |
| 7 | STA | TISTICAL METHODOLOGY AND STATISTICAL ANALYSES | 6 |
| | 7.1 | STATISTICAL METHODS | 6 |
| | 7.2 | STATISTICAL ANALYSES | 7 |
| | 7.2.1 | ! Safety Analysis | 7 |
| | 7.2.2 | , | |
| | 7.2.3 | | |
| | | Analyses of Secondary Endpoint | |
| | | 5 Summary of Analyses | |
| 8 | LIS | T OF LISTINGS AND TABLES | 15 |
| 9 | REF | FERENCES | 16 |
| 1( | 0 APP | PENDICES | 17 |
| | 10.1 | APPENDIX 1: MOCK SHELLS FOR TABLES | 17 |
| | 10.2 | APPENDIX 2: MOCK SHELLS FOR LISTINGS | 17 |
| | | PEIZER CONFIDENTIAL | |

### 1 AMENDMENTS FROM PREVIOUS VERSION(S)

Not Applicable

#### 2 INTRODUCTION

This is a non-interventional retrospective study to examine the real world usage, effectiveness, and safety of ceftazidime-avibactam for the treatment of Gram negative infections in India. 500 hospitalized patients who have received at least 48 hours of Ceftazidime- Avibactam. Data will be collected for the period of 01 June 2019 till 01 April 2020. The patient should have completed treatment with ceftazidime-avibactam before 01 April 2020. The data collection will stop once data from 500 patients has been abstracted

This statistical analysis plan (SAP) will be the guiding document for the analyses that will be conducted in the study. We intend to understand the real world usage, efficacy and safety of Ceftazidime avibactam in treating Gram negative infections. SAP describes the data to be summarized and analyzed, including specifics of the statistical analyses to be performed.

This statistical analysis plan (SAP) is based on protocol version 2.0 dated 21st October 2020 and case report form (CRF) version 4 Jan 2021.

#### 2.1 STUDY DESIGN

This is a non-interventional retrospective study to examine the real-world usage, effectiveness, and safety of ceftazidime-avibactam for the treatment of gram-negative infections in India. 500 hospitalized patients who have received at least 48 hours of Ceftazidime- Avibactam. Data will be collected for the period of 01 June 2019 till 01 April 2020. The patient should have completed treatment with ceftazidime-avibactam before 01 April 2020. The data collection will stop once data from 500 patients has been abstracted.

Data will be collected through the abstraction of hospital medical records (electronic) if available or through the individual patient case files (paper) in case electronic records are not available. Collected study data will include but will not be limited to patient characteristics, clinical and microbiologic characteristics of the infection, and treatment patterns, effectiveness, and safety of ceftazidime-avibactam.

#### Study population

All hospitalized patients who have received at least 48 hours of ceftazidime-avibactam

### Data source

Data from the patients who have received Ceftazidime-Avibactam as a part of the routine clinical management for Gram negative infections will be recorded as per the defined outcomes. Data will be abstracted from electronic health records. Individual patient medical records, in case is necessary. The data will be abstracted by a CRO (clinical

research organization), the principal investigator (PI) or a reviewer (clinical research associate) nominated by the PI. For the records missing any of the requested information, data will be reported as missing. Data from patients that were part of the named access program will be excluded.

### **Treatment/cohort labels**

Ceftazidime-avibactam

#### 2.2 STUDY OBJECTIVES

### Primary Objective:

- Describe the treatment success of patients treated with ceftazidime-avibactam at Day 7, Day 14/ end of treatment after ceftazidime-avibactam initiation, whichever is earlier.
- 2. Describe the microbiological success among patients treated with ceftazidimeavibactam at day 7, Day 14/ end of treatment after Ceftazidime avibactam initiation whichever is earlier.
- 3. Number of patients with serious and non-serious AEs with explicit attribution to Ceftazidime avibactam for up to 30 days post treatment completion with Ceftazidime-Avibactam, death or discharge; whatever is first.

### Secondary Objective:

- 1. Describe the source of infection at baseline for which ceftazidime-avibactam was used.
- 2. Describe the indications and reasons for use of ceftazidime-avibactam at baseline.
- 3. Describe the dose in mg, frequency of dose in hours, duration in days, and combination antibiotic regimen given till 14 days/ End of treatment whichever is earlier.
- 4. Describe at baseline any prior antimicrobial therapy administered in the 90 days prior to current admission.
- 5. Describe the gram-negative organisms identified and the susceptibility to ceftazidime avibactam along with molecular typing at baseline.
- 6. Describe the in-hospital length of stay (LOS) in days, LOS in ICU in days and percentage of various healthcare resource utilization in patients with infections treated by ceftazidime-avibactam up to 30 days post treatment completion with Ceftazidime-Avibactam death or discharge; whatever is first.
- 7. Determine the incidence of recurrent infections during the hospital stay, including re-infection and relapse up to 30 days post treatment completion with Ceftazidime-Avibactam, death or discharge; whatever is first.

#### 3 HYPOTHESES AND DECISION RULES

#### 3.1 STATISTICAL HYPOTHESES

Not Applicable

#### 3.2 STATISTICAL DECISION RULES

Not Applicable

#### 4 ANALYSIS SETS/POPULATIONS

#### 4.1 ALL SUBJECTS SET

All available data from all subjects who have received at least 48 hours (or three doses) of Ceftazidime- Avibactam will be used for summary/analysis purpose

#### 4.2 SAFETY ANALYSIS SET

The safety analysis set is the same as the all subjects set.

#### 4.3 OTHER ANALYSIS SET

Not Applicable

### 4.4 SUBGROUPS

Not Applicable

#### 5 ENDPOINTS AND COVARIATES

### 5.1 EFFICACY/EFFECTIVENESS ENDPOINT(S)

- Treatment success of patients treated with ceftazidime-avibactam at Day 7, Day 14/ end of treatment after ceftazidime-avibactam initiation, whichever is earlier.
- Microbiological success among patients treated with ceftazidime-avibactam at day 7, Day 14/ end of treatment after Ceftazidime avibactam initiation whichever is earlier.
- Source of infection at baseline for which ceftazidime-avibactam was used.
- Indications and reasons for use of ceftazidime-avibactam at baseline
- Dose in mg, frequency of dose in hours, duration in days, and combination antibiotic regimen given till 14 days/ End of treatment whichever is earlier.
- Any prior antimicrobial therapy administered in the 90 days prior to current admission.
- The gram-negative organisms identified and the susceptibility to ceftazidime avibactam along with molecular typing at baseline.
- The in-hospital length of stay (LOS) in days, LOS in ICU in days and percentage
  of various healthcare resource utilization in patients with infections treated by
  ceftazidime-avibactam up to 30 days post treatment completion with CeftazidimeAvibactam death or discharge; whatever is first.

#### 5.2 SAFETY ENDPOINTS

 Number of patients with serious and non-serious AEs with explicit attribution to Ceftazidime avibactam for up to 30 days post treatment completion with Ceftazidime- Avibactam, death or discharge; whatever is first.

• incidence of recurrent infections during the hospital stay, including re-infection and relapse up to 30 days post treatment completion with Ceftazidime-Avibactam, death or discharge; whatever is first.

#### 5.3 OTHER ENDPOINTS

Not Applicable

### 5.4 COVARIATES

Not Applicable

#### 6 HANDLING OF MISSING VALUES

No imputation for missing values will be performed.

#### 7 STATISTICAL METHODOLOGY AND STATISTICAL ANALYSES

#### 7.1 STATISTICAL METHODS

Analysis of the data will be performed by the Biostatistics and Statistical Programming team. All statistical analyses will be performed using SAS® Version 9.4 or higher [SAS Institute Inc., USA]. The SAP will be finalized before database lock.

The following standard descriptive summaries will be presented:

#### Descriptive statistics for continuous data:

The continuous data will be summarized using the number of observations (n), arithmetic mean (mean), standard deviation (SD), median, minimum value (min), and maximum value (max).

The number of observations (n) will be presented with no decimal place, mean and median will be presented up to one decimal place from the original value, SD up to two decimal places from the original value and (min, max) as an original value.

#### Descriptive statistics for categorical data:

The categorical variables will be summarized using the frequency count (n) and percentage (%) for each possible value. The frequencies will be presented up to 0 decimal places, percentage up to 1 decimal place.

If data are not available, a missing category will be presented. Statistical tests, if any, will be performed at 5% level of significance. The denominator for percentages will be based on the number of patients appropriate for the purpose of the analysis.

#### 7.2 STATISTICAL ANALYSES

### 7.2.1 Safety Analysis

#### • Adverse Events

Any signs, symptoms, illnesses or diagnosis (either observed or volunteered) that appear or worsen during the course of the study are recorded as Adverse Events.

Adverse events with explicit attribution to any Pfizer drug that appear in the reviewed information (defined per the patient population and study period specified in the protocol) will be reported. Explicit attribution is not inferred by temporal relationship between drug administration and an AE, but must be based on a definite statement of causality by a healthcare provider linking drug administration to the AE.

The requirements for reporting safety events on the non-interventional study (NIS) adverse event monitoring (AEM) Report Form to Pfizer Safety are as follows:

- All serious and non-serious AEs with explicit attribution to any Pfizer drug that appear in the reviewed information must be recorded on the Case record form and reported, within 24 hours of awareness, to Pfizer Safety using the NIS AEM Report Form.
- O Scenarios involving drug exposure, including exposure during pregnancy, exposure during breast feeding, medication error, overdose, misuse, extravasations, lack of efficacy, and occupational exposure associated with the use of a Pfizer product must be reported, within 24 hours of awareness, to Pfizer Safety using the NIS AEM Report Form.

### • Serious Adverse Event (SAE)

Serious adverse event is defined as an event that meets any one of the criteria given below.

- Life threatening (in the opinion of the investigator, the subject is at immediate risk of death from the event [substantial risk of dying at the time of the adverse event])
- A persistent or significant disability/incapacity (a substantial disruption of a person's ability to conduct normal life functions)
- o Fatal
- o Requires or Prolongs Hospitalization
- o Congenital anomaly or birth defect
- o Other medically important adverse events.

#### Non-serious Adverse Event

All AEs that do not meet the criteria for "serious" are considered as non-serious.

### Relationship

The relationship of each AE to drug will be classified as below.

- o Adverse event related to ceftazidime-avibactam
- o Adverse event related to concomitant drug
- o Adverse event related to other Pfizer drug

#### Analysis of Adverse Events

All the adverse events (AEs )and serious adverse events (SAEs) reported throughout the study shall be coded and classified along the standards of MedDRA (Medical Dictionary for Regulatory Activities) version 23.0 and grouped by preferred term (PT) and system organ class (SOC).

Subject counts (n) and percentages (%) will be presented for all the subjects. If a subject has more than one AE, subject will be counted only once in SOC and once for each PT. If a subject has more than one episode of an AE, the subject will be counted only once within a specific preferred term. Number of subjects with event (n) and the percentage of subjects exposed to event (%) will be tabulated.

Summarization for AEs by subjects will be provided for following categories:

- o All Adverse Events
- o AE's By SOC And PT
- o Serious AEs by SOC and PT
- o Drug Related AEs by SOC and PT
- o AEs leading to death by SOC and PT
- o AEs leading to permanent discontinuation
- o AE's By SOC, PT And Severity
- o Drug Related AEs by SOC and PT and Severity

#### Additional risk factor

The additional risk factor data will be summarized at each visit using frequencies (n) and percentages (%) for safety population.

### • Laboratory Investigations

The Microbiology and pathogen susceptibility data will be summarized using descriptive statistics and frequency count and percentage of each pathogen organism.

Pathogen susceptibility: All susceptibility information will be collected for the isolated pathogens including tested antibiotic by classes (e.g. aminoglycosides, amphenicol, beta-lactams, carbapenems, cephalosporins, glycopeptides, glycylcyclines, lipopeptides, macrolides, monobactams, nitroimidazoles, oxazolidinones, penicillins, penicillins and beta-lactamase inhibitors, quinolones, streptogramins, tetracyclines, other) and within class, and sensitivity to each (susceptible, intermediate, resistant).

### 7.2.2 Subjects and Site Characteristics

#### • Site Characteristics

Medical specialty of the treating physician indicating Ceftazidime- Avibactam (e.g. infectious disease, surgical). Care level, Hospital type, number of beds, number of ICU beds will be summarized using by frequency (n) and percentage (%).

### • Local Gram-Negative Resistance Patterns

Multidrug-resistance: The isolate is non-susceptible to at least 1 agent in  $\geq 3$  antimicrobial categories. Categories include but are not limited to aminoglycosides, carbapenems, cephalosporins, cephamycins, fluoroquinolones, folate pathway inhibitors, glycylcyclines, penicillins, monobactams, phosphonic acids, polymyxins, tetracyclines.

Any hospitalized adult patient with an infection caused by known gram negative pathogens at baseline will be categorized and presented by frequency (n) and percentage (%). The rate (%) available for percentage of gram-negative isolates that exhibit resistance to 3rd generation drugs (cephalosporins, carbapenem, cephalosporins and carbapenem, colistin) will be summarized using descriptive statistics.

### • Demographic Characteristics

The demographic and baseline characteristics will be summarized by using descriptive statistics. Continuous variables such as age, height, weight, will be summarized by number of observations (n), arithmetic mean (mean), standard deviation (SD), median, minimum value (min), and maximum value (max) and Categorical variables such as gender, race, Current employment status, will be presented by frequency (n) and percentage (%).

#### Index Hospitalization

Details of index hospitalization such as mode of admission, source of admission, ward admitted for initial hospitalization, diagnosis and current admission to ICU will be summarized by frequency (n) and percentage (%).

#### Additional Risk Factors

Additional risk factors such as patient travelled to any foreign country in last 3 months, pregnancy, alcohol use, tobacco use will be summarized by frequency (n) and percentage (%).

### • Prior and Concomitant Antibiotic Therapy

For all prior antibiotics(s), prior lines of treatment (Antibiotic(s)) used for current infection before ceftazidime-avibactam initiation, antibiotics(s) used concurrently with ceftazidime-avibactam, frequency counts (n) & percentages (%) of patients will be presented by verbatim terms and will be sorted in descending order of frequency.

#### • Antibiotic Treatment After Ceftazidime-Avibactam

For all antibiotics treatment after Ceftazidime-Avibactam, frequency counts (n) & percentages (%) of patients will be presented by verbatim terms and will be sorted in descending order of frequency.

#### Renal Status of Patient

Any patients with renal dysfunction will be presented by frequency (n) and percentage (%). Renal parameters such as serum creatinine and CRCL will be summarized using descriptive statistics and severity of renal dysfunction will be summarized by frequency (n) and percentage (%).

#### • Recent hospitalization and healthcare procedure

Recent hospitalization and healthcare procedure will be listed only.

Hospital stay and healthcare utilization (diagnosis at admission, departments admitted/discharged, discharge diagnosis, mechanical ventilation, dialysis, CT/MRI imaging, tracheotomy, surgical intervention, and percutaneous procedures) will be summarized using frequency count (n) and percentage (%) of patients for the safety population.

### • Comorbidities (DEYO-CHARLSON COMORBIDITY INDEX)

For all comorbidities, frequency counts (n) & percentages (%) of patients will be presented. The Deyo-Charlson Comorbidity Index (DCCI) will be used to predict patients' 10-year probability of survival and will be used as a measure of overall health. The comorbidities evaluated in the DCCI will be collected at baseline from medical records to calculate the score. The DCCI Score will be summarized using the descriptive statistics (n, mean, SD, minimum and maximum).

#### 7.2.3 Analyses of Primary Endpoint

• Treatment success of patients treated with ceftazidime-avibactam at Day 7, Day 14/ end of treatment after ceftazidime-avibactam initiation, whichever is earlier.

The clinical symptom improvement will be assessed as symptom improved, symptom worsened, and not assessed and summarized by frequency count (n) and percentage (%) at 72hrs (Day3), Day 7 and Day 14/ end of treatment.

The treatment success is defined as resolution of all signs and symptoms of the infection. This will be as per the clinician's judgment and the treatment protocol/algorithm followed at the respective centers. The treatment success in terms of clinical outcome classified mainly in three groups, clinical success, clinical failure and indeterminate of patients treated with ceftazidime-avibactam and will be summarized in terms of frequency count (n) and percentage (%) at Day 7 and Day 14/ end of treatment after ceftazidime-avibactam initiation, whichever is earlier.

 Microbiological success among patients treated with ceftazidime-avibactam at day 7, Day 14/ end of treatment after Ceftazidime-avibactam initiation whichever is earlier.

The microbiological success defined as absence of causative pathogen from appropriately obtained specimens at the site of infection (Eradication) and repeat cultures were not performed/clinically indicated in a patient who had a clinical response of cure (Presumed Eradication).

The microbiological outcomes are classified as microbiological success and failure and will be summarized by frequency count (n) and percentage (%) at Day 7 and Day 14/ end of treatment after ceftazidime-avibactam initiation, whichever is earlier.

 Number of patients with serious and non-serious AEs with explicit attribution to Ceftazidime-avibactam for up to 30 days post treatment completion with Ceftazidime- Avibactam, death or discharge; whatever is first.

Details of adverse event analysis is provided in section 7.2.1

### 7.2.4 Analyses of Secondary Endpoint

Source of infection at baseline for which ceftazidime-avibactam was used.

Source of infection includes hospital-acquired infection (HAI) healthcareassociated infection (HCAI), and community-acquired infection (CAI). The source of infection at baseline will be summarized using the frequency count (n) and percentage (%) for each source of infection.

Indications and reasons for use of ceftazidime-avibactam at baseline.

The indications and reasons for use of ceftazidime-avibactam at baseline includes UTI, IAI, NP and any other indication with its reasons such as primary diagnosis, secondary diagnosis, symptoms etc will be summarized using the frequency count (n) and percentage (%) for each possible value.

 Description of dose in mg, frequency of dose in hours, duration in days, and combination antibiotic regimen given till 14 days/ End of treatment whichever is earlier.

Proportion of patients with use of ceftazidime-avibactam for >=48 hours reported in patient records will be summarized using frequency counts (n) & percentages (%).

The dose in mg, duration of administration and total duration of therapy of ceftazidime - avibactam exposure will be summarized by number of observations (n), arithmetic mean (mean), standard deviation (SD), median, minimum value (min), and maximum value (max) till 14 days/ End of treatment whichever is earlier. Frequency of dose, category of treatment, reason for discontinuation will be summarized using frequency counts (n) & percentages (%) of patients till 14 days/ End of treatment whichever is earlier.

For all combination of antibiotic regimen, a table of concomitant antibiotic therapy will be provided as per section 7.2.2

 Any prior antimicrobial therapy administered in the 90 days prior to current admission at baseline.

Any prior antimicrobial therapy administered in the 90 days prior to current admission will be presented in the table of History of Prior Antibiotic Exposure as per section 7.2.2

 Describe the gram-negative organisms identified and the susceptibility to ceftazidime -avibactam along with molecular typing at baseline.

The gram-negative organisms identified and susceptibility to ceftazidime - avibactam at baseline will be summarized using frequency counts (n) & percentages (%).

• Describe the in-hospital length of stay (LOS) in days, LOS in ICU in days and percentage of various healthcare resource utilization in patients with PFIZER CONFIDENTIAL

Page 12 of 17

infections treated by ceftazidime-avibactam up to 30 days post treatment completion with Ceftazidime- Avibactam death or discharge; whatever is first.

The in-hospital length of stay (LOS) in days will be calculated based on 1) total number of consecutive days the patient was treated in the hospital from admission to discharge during their initial hospitalization; 2) the total number of days hospitalization between diagnosis of infection and discharge; 3) the total number of days the patient was treated in the hospital after ceftazidime-avibactam initiation up to hospital discharge, including the first day of treatment.

ICU LOS will be calculated as: 1) the total number of consecutive or non-consecutive days the patient was treated in the ICU during their initial hospitalization; and 2) the total number of days the patient was treated in the ICU after ceftazidime-avibactam initiation, including the first day of treatment.

The in-hospital length of stay (LOS) in days, LOS in ICU in days with infections treated by ceftazidime-avibactam up to 30 days post treatment completion with Ceftazidime- Avibactam death or discharge; whatever is first will be summarized using the number of observations (n), arithmetic mean (mean), standard deviation (SD), median, minimum value (min), and maximum value (max)

Healthcare resource utilization data (medical/surgical/percutaneous procedures, CT/MRI imaging, days of mechanical ventilation, days of dialysis) will be abstracted from the patient medical records and summarize using frequency counts (n) & percentages (%).

• Incidence of recurrent infections during the hospital stay, including reinfection and relapse up to 30 days post treatment completion with Ceftazidime- Avibactam, death or discharge; whatever is first.

Any incidence of recurrent infections during the hospital stays, including reinfection and relapse up to 30 days post treatment completion with Ceftazidime-Avibactam, death or discharge; whatever is first will be summarized using frequency counts (n) & percentages (%) of patients will be presented by verbatim terms and will be sorted in descending order of frequency.

7.2.5 Summary of Analyses

#### Outcome Analysis Set Supports Subgroup Statistical Method Missing Data Covariates/Strata Protocol **Primary** Objective Number Frequency count (n) and All Subjects Set Not Applicable Not Applicable Excluded Treatment success 1 percentage (%) Frequency count (n) and Microbiological success All Subjects Set 2 Not Applicable Not Applicable Excluded percentage (%) Number of patients with Frequency count (n) and All Subjects Set Not Applicable 3 Not Applicable Excluded serious and non-serious AEs percentage (%)

#### 8 LIST OF LISTINGS AND TABLES

- Listing 16.2.1.1 Site Characteristics- All subjects data
- Listing 16.2.1.2 Local Gram-negative Resistance Patterns All Subjects Data
- Listing 16.2.1.3 Demographic Characteristics Safety Population
- Listing 16.2.2.1 Renal Status of Patient Safety Population
- Listing 16.2.2.2 Comorbidities (Deyo-Charlson Comorbidity Index) All Subjects
- Listing 16.2.2.3 Disease Severity All Subjects
- Listing 16.2.2.4 Additional Risk Factor -All Subjects
- Listing 16.2.3.1 Index Hospitalization -All Subjects
- Listing 16.2.3.2 Length of Hospital Stay Safety Population
- Listing 16.2.3.3 Current Admission to ICU All Subjects
- Listing 16.2.3.4 Prior Recent Hospitalization -Safety Population
- Listing 16.2.3.5 Recent Healthcare Procedures -Safety Population
- Listing 16.2.3.6 Healthcare Utilization Safety Population
- Listing 16.2.4.1 Indication All Subjects
- Listing 16.2.5.1 Ceftazidime-Avibactam Exposure All Subjects
- Listing 16.2.5.2 History of Prior Antibiotic Exposure All Subject Data
- Listing 16.2.5.3 Concomitant Antibiotic Therapy All Subject Data
- Listing 16.2.5.4 Antibiotic Therapy: Prior lines of Treatment All Subjects
- Listing 16.2.5.5 Antibiotic Treatment After Ceftazidime-Avibactam All Subjects
- Listing 16.2.6.1 Clinical Symptoms Improvement– All Subjects
- Listing 16.2.6.2 Microbiological Evaluation Safety Population
- Listing 16.2.6.3 Recurrence of Infection Safety Population
- Listing 16.2.6.4 Susceptibility to Ceftazidime-Avibactam All Subjects
- Listing 16.2.7.1 Microbiology- All Subjects
- Listing 16.2.7.2 Pathogen Susceptibility Safety Population
- Listing 16.2.8.1 In-Hospital Mortality Safety Population
- Listing 16.2.9.1 Adverse Events Safety Population
- Table 14.1.1.1 Site Characteristics All Subjects
- Table 14.1.1.2 Local Gram-Negative Resistance Patterns-All Subjects
- Table 14.1.2.1 Demographic Characteristics All Subjects
- Table 14.1.2.2 Index Hospitalization All Subjects
- Table 14.1.2.3 Additional Risk Factors All Subjects
- Table 14.1.2.4 History of Prior Antibiotic Exposure –All Subjects
- Table 14.1.2.5 Concomitant Antibiotic Therapy–All Subjects
- Table 14.1.2.6 Antibiotic Therapy: Prior Lines of Treatment -All Subject
- Table 14.1.2.7 Antibiotic treatment after Ceftazidime-Avibactam –All Subjects
- Table 14.1.2.8 Renal Status of Patient All Subjects

- Table 14.1.2.9 Comorbidities (Deyo-Charlson Comorbidity Index) -All Subjects
- Table 14.1.2.10 Indwelling Devices at the time of Infection Diagnosis All Subejcts
- Table 14.1.2.11 Disease Severity -All Subjects
- Table 14.1.2.12 Source of Infection at Baseline All Subjects
- Table 14.1.2.13 Indications and Reasons for Use of Ceftazidime-Avibactam- All Subjects
- Table 14.2.1.1 Clinical Symptom Improvement –All Subjects
- Table 14.2.1.2 Microbiological Evaluation -All Subjects
- Table 14.2.2.3 Gram Negative Organisms Identified All Subjects
- Table 14.2.2.4 Susceptibility to Ceftazidime -Avibactam All Subjects
- Table 14.2.2.5 Length of Stay in Hospital/ICU All Subjects
- Table 14.3.1.1 Ceftazidime Avibactam Exposure- All Subjects
- Table 14.3.2.1 Summary of Subjects with AEs -All Subjects
- Table 14.3.2.2 Summary of Subjects With AE's by Soc And PT- All Subjects
- Table 14.3.2.3 Summary of Subjects with Serious AEs by SOC and PT All Subjects
- Table 14.3.2.4 Summary of Subjects with Study Drug Related AEs by SOC and PT All Subjects
- Table 14.3.2.5 Summary of Subjects with other Pfizer Drug Related AEs by SOC and PT All Subjects
- Table 14.3.2.6 Summary of Subjects with AEs leading to death by SOC and PT All Subjects
- Table 14.3.2.7 Summary of Subjects with AEs leading to permanent discontinuation of study drug by SOC and PT -All Subjects
- Table 14.3.3.1 Recurrence of Infection All Subjects
- Table 14.3.4.1 Microbiology Results- All Subjects
- Table 14.3.5.1 Pathogen Susceptibility All Subjects
- Table 14.3.6.1 In-Hospital Mortality All Subjects

### 9 REFERENCES

- 1. X9001260, Version 2.0, October 20, 2020
- 2. X9001260, CRF Version, January 4, 2021

### 10 APPENDICES

- 10.1 APPENDIX 1: MOCK SHELLS FOR TABLES
- 10.2 APPENDIX 2: MOCK SHELLS FOR LISTINGS

Protocol Number: X9001260 Status=SHELLS Page X of Y

Program Name: Txx.sas Produced: DDMMMYYYY

#### **Appendix 10.1 Mock Shells for Tables**

#### General Notes for programmers:

1. For more details regarding tables please refer to SAP write-up, protocol, CRF and metadata.

2. If there are no counts in any of the tables then display the line "No Subject Meets the Reporting Criteria" in the body of tables.

3. First two title on each table is as follows

Protocol Number: X9001260 Status=SHELLS Page X of Y

Program Name: Txx.sas Produced: DDMMMYYYY

Where Status of the report should be Shells (at Draft stage) and change to Final (for Final output). Please refer to first table

- 4. Report should be produced with "Times New Roman" as text font and height of the text should be 9.
- 5. Report should have Left, Right, Top and Bottom Margins to 1.
- 6. Footnote text mentioned in Mock Shell starts with "Programmer's Note: " is only a note for Programmer and is not a part of Report.
- 7. Footnote text mentioned in Mock Shell starts with "Note" will be presented as footnote during generation of tables.

Program Name: Txx.sas

Produced: DDMMMYYYY

Page X of Y

### Table of Content

| Table 14.1.1.1 Site Characteristics – All Subjects | ∠ |
|---|---|
| Table 14.1.1.2 Local Gram-Negative Resistance Patterns-All Subjects | 6 |
| Table 14.1.2.1 Demographic Characteristics – All Subjects | 8 |
| Table 14.1.2.2 Index Hospitalization – All Subjects | |
| Table 14.1.2.3 Additional Risk Factors – All Subjects | 10 |
| Table 14.1.2.4 History of Prior Antibiotic Exposure –All Subjects | 11 |
| Table 14.1.2.5 Concomitant Antibiotic Therapy–All Subjects | 11 |
| Table 14.1.2.6 Antibiotic Therapy: Prior Lines of Treatment –All Subject | 11 |
| Table 14.1.2.7 Antibiotic treatment after Ceftazidime-Avibactam –All Subjects | 11 |
| Table 14.1.2.8 Renal Status of Patient – All Subjects | 12 |
| Table 14.1.2.9 Comorbidities (Deyo-Charlson Comorbidity Index) –All Subjects | 13 |
| Table 14.1.2.10 Indwelling Devices at the time of Infection Diagnosis – All Subejcts | 14 |
| Table 14.1.2.11 Disease Severity –All Subjects | 15 |
| Table 14.1.2.12 Source of Infection at Baseline – All Subjects | 16 |
| Table 14.1.2.13 Indications and Reasons for Use of Ceftazidime-Avibactam– All Subjects | 17 |
| Table 14.2.1.1 Clinical Symptom Improvement –All Subjects | 18 |
| Table 14.2.1.2 Microbiological Evalustion –All Subjects | 19 |

| Table 14.2.2.3 Gram Negative Organisms Identified – All Subjects | 20 |
|---|---|
| Table 14.2.2.4 Susceptibility to Ceftazidime -Avibactam – All Subjects | 22 |
| Table 14.2.2.5 Length of Stay in Hospital/ICU – All Subjects | 22 |
| Table 14.3.1.1 Ceftazidime - Avibactam Exposure - All Subjects | 23 |
| Table 14.3.2.1 Summary of Subjects with AEs –All Subjects | 25 |
| Table 14.3.2.2 Summary of Subjects With AE's by Soc And PT- All Subjects | 27 |
| Table 14.3.2.3 Summary of Subjects with Serious AEs by SOC and PT – All Subjects | 27 |
| Table 14.3.2.4 Summary of Subjects with Study Drug Related AEs by SOC and PT – All Subjects | 27 |
| Table 14.3.2.5 Summary of Subjects with other Pfizer Drug Related AEs by SOC and PT – All Subjects | 27 |
| Table 14.3.2.6 Summary of Subjects with AEs leading to death by SOC and PT – All Subjects | 27 |
| Table 14.3.2.7 Summary of Subjects with AEs leading to permanent discontinuation of study drug by SOC and PT -All Subjects | 27 |
| Table 14.3.3.1 Recurrence of Infection – All Subjects | 28 |
| Table 14.3.4.1 Microbiology Results– All Subjects | 29 |
| Table 14.3.5.1 Pathogen Susceptibility – All Subjects | 30 |
| Table 14.3.6.1 In-Hospital Mortality – All Subjects | 32 |

Table 14.1.1.1 Site Characteristics – All Subjects

| Characteristic (Unit) | Statistics | Ceftazidime-avibactam |
|-----------------------|------------|-----------------------|
| | | (N = xx) |
| Di ii a iii | | |
| Physician Speciality | | |
| Infectious disease | n (%) | xx(xxx) |
| Microbiology | n (%) | xx(xxx) |
| Surgical | n (%) | xx(xxx) |
| Internal medicine | n (%) | xx(xxx) |
| Intensive care | n (%) | xx(xxx) |
| Anesthesiology | n (%) | xx (xx x) |
| Other (specify) | n (%) | xx (xx x) |
| Hospital Information | | |
| Care Level | | |
| Secondary | n (%) | xx(xxx) |
| Tertiary | n (%) | xx (xx x) |
| Hospital Type | | |
| Teaching | n (%) | xx (xx x) |
| Non-Teaching | n (%) | xx (xx x) |
| Total no. of Beds | n | XX |
| | Mean (SD) | xx x(xx xx) |
| | Median | xx x |
| | Min, Max | xx, xx |
| Total no. of ICU Beds | n | XX |
| | Mean (SD) | xx x(xx xx) |
| | Median | xx x |
| | Min, Max | xx, xx |

Protocol Number: X9001260 Status=SHELLS Page X of Y

Program Name: Txx.sas Produced: DDMMMYYYY

Abbreviations: N = number of subjects in Ceftazidime-avibactam group; n = number of subjects in specified category

Note 1: Percentages are based on the number of subjects in the Ceftazidime-avibactam group.

Table 14.1.1.2 Local Gram-Negative Resistance Patterns-All Subjects

| Characteristic (Unit) | Statistics | Ceftazidime-avibactam $(N = xx)$ |
|---|---|---|
| Percentage of gram-negative isolates that exhibit resistance to 3rd generation known for | | |
| Cephalosporins | | |
| Yes | n (%) | xx (xx x) |
| No | n (%) | xx (xx x) |
| Cephalosporins Rate | n | XX |
| | Mean (SD) | xx x(xx xx) |
| | Median | xx x |
| | Min, Max | xx, xx |
| Carbapenem | | |
| Yes | n (%) | xx (xx x) |
| No | n (%) | xx (xx x) |
| Carbapenem Rate | n | xx |
| | Mean (SD) | xx x(xx xx) |
| | Median | xx x |
| | Min, Max | xx, xx |
| Cephalosporins and Carbapenem | | |
| Yes | n (%) | xx (xx x) |
| No | n (%) | xx(xxx) |
| Cephalosporins and Carbapenem Rate | n | XX |
| | Mean (SD) | xx x(xx xx) |
| | Median | XX X |
| | Min, Max | xx, xx |

| Colistin | | |
|---------------|-----------|-------------|
| Yes | n (%) | xx (xx x) |
| No | n (%) | xx (xx x) |
| Colistin Rate | n | xx |
| | Mean (SD) | xx x(xx xx) |
| | Median | XX X |
| | Min, Max | xx, xx |

Abbreviations: N = number of subjects in Ceftazidime-avibactam group; n = number of subjects in specified category

Note 1: Percentages are based on the number of subjects in the Ceftazidime-avibactam group. Reference listing xxxxxx

Table 14.1.2.1 Demographic Characteristics – All Subjects

| Characteristic (Unit) | Statistics | Ceftazidime-avibactam $(N = xx)$ |
|---------------------------|------------|----------------------------------|
| Gender | | |
| Male | n (%) | xx (xx x) |
| Female | n (%) | xx(xxx) |
| Age (Years) | n | XX |
| | Mean (SD) | xx x(xx xx) |
| | Median | XX X |
| | Min, Max | XX, XX |
| Height (cm) | n | XX |
| | Mean (SD) | xx x(xx xx) |
| | Median | XX X |
| | Min, Max | XX, XX |
| Weight (cm) | n | XX |
| | Mean (SD) | xx x(xx xx) |
| | Median | XX X |
| | Min, Max | XX, XX |
| Current employment status | | |
| Full Time | n (%) | xx (xx x) |
| Part Time | n (%) | xx (xx x) |
| Unemployed | n (%) | xx (xx x) |
| Retired | n (%) | xx (xx x) |
| Not Applicable | n (%) | xx (xx x) |

Abbreviations: N = number of subjects in Ceftazidime-avibactam group; n = number of subjects in specified category Note 1: Percentages are based on the number of subjects in the Ceftazidime-avibactam group.

Reference listing xxxxxx

Table 14.1.2.2 Index Hospitalization – All Subjects

| Characteristic (Unit) | Statistics | Ceftazidime-avibactam |
|---|---|---|
| | | (N = xx) |
| Mode of admission | | |
| Emergency | n (%) | xx (xx x) |
| Scheduled | n (%) | xx (xx x) |
| Source of admission | | |
| Outpatient | n (%) | xx (xx x) |
| Long term care facility | n (%) | xx (xx x) |
| Transfer from acute care hospital | n (%) | xx (xx x) |
| Direct Admission | n (%) | xx (xx x) |
| Other | n (%) | xx (xx x) |
| Ward admitted for initial hospitalization | | |
| Surgical | n (%) | xx (xx x) |
| Medical | n (%) | xx (xx x) |
| Onco-hematology | n (%) | xx (xx x) |
| Infectious disease | n (%) | xx (xx x) |
| ICU | n (%) | xx (xx x) |
| Other | n (%) | xx (xx x) |
| Current admission to ICU | | |
| Yes | n (%) | xx (xx x) |
| No | n (%) | xx (xx x) |

Abbreviations: N = number of subjects in Ceftazidime-avibactam group; n = number of subjects in specified category Note 1: Percentages are based on the number of subjects in the Ceftazidime-avibactam group.

Reference listing xxxxxx

Table 14.1.2.3 Additional Risk Factors – All Subjects

| Characteristic (Unit) | Statistics | Ceftazidime-avibactam $(N = xx)$ |
|---|---|---|
| Patient Travelled to any foreign country in t | he last 3 months | |
| Yes | n (%) | xx (xx x) |
| No | n (%) | xx (xx x) |
| Pregnancy | | |
| Yes | n (%) | xx (xx x) |
| No | n (%) | xx (xx x) |
| Not Applicable | n (%) | xx (xx x) |
| Alcohol Use | | |
| Yes | n (%) | xx (xx x) |
| No | n (%) | xx (xx x) |
| Unknown | n (%) | xx (xx x) |
| Tobacco Use | | |
| Current Smoker | n (%) | xx (xx x) |
| Previous Smoker | n (%) | xx (xx x) |
| Never Smoked | n (%) | xx (xx x) |
| Unknown | n (%) | xx (xx x) |

Abbreviations: N = number of subjects in Ceftazidime-avibactam group; n = number of subjects in specified category Note 1: Percentages are based on the number of subjects in the Ceftazidime-avibactam group.

Reference listing xxxxxx

Table 14.1.2.4 History of Prior Antibiotic Exposure –All Subjects

| Generic Drug Name | Statistics | Ceftazidime-<br>avibactam<br>(N = xx) |
|---|---|---|
| Number of Subjects with at Least One Prior Antibiotic Medication | n(%) | xx ( xx x) |
| XXXXXXX | n(%) | xx (xx.x) |
| XXXXXXX | n(%) | xx (xx.x) |
| XXXXXXX | n(%) | xx (xx x) |

Abbreviations: N = number of subjects in Ceftazidime-avibactam; n = number of subjects in specified category

Note 1: Percentages are based on number of subjects in Ceftazidime-avibactam group

Reference Listing xxxxx

Programmer's Note 1: The above table will be continued for other ATC texts.

Programmers Note: ATC level 2 texts and Generic Name will be sorted in descending order of frequency.

Similar table will be presented as follows:

Table 14.1.2.5 Concomitant Antibiotic Therapy—All Subjects
Table 14.1.2.6 Antibiotic Therapy: Prior Lines of Treatment –All Subject
Table 14.1.2.7 Antibiotic treatment after Ceftazidime-Avibactam –All Subjects

Table 14.1.2.8 Renal Status of Patient – All Subjects

| Test(Unit) | Statistics | Ceftazidime-avibactam |
|--------------------------|------------|-----------------------|
| | | (N = xx) |
| Renal dysfunction | | |
| Yes | n(%) | xx(xx x) |
| No | n(%) | xx(xx x) |
| Serum Creatinine (mg/dl) | N | XX |
| | Mean (SD) | xx x (xx xx) |
| | Median | xx x |
| | Min, Max | XX, XX |
| CRCL(ml/min) | N | XX |
| | Mean (SD) | xx x (xx xx) |
| | Median | XX X |
| | Min, Max | XX, XX |
| Renal dysfunction | | |
| Mild | n(%) | xx(xx x) |
| Moderate | n(%) | xx(xx x) |
| Severe | n(%) | xx(xx x) |

Abbreviations: N = number of subjects in Ceftazidime-avibactam group; n = Number of subjects in specified category. Reference Listing xxxxxx

Table 14.1.2.9 Comorbidities (Deyo-Charlson Comorbidity Index) – All Subjects

| Characteristic (Unit) | Statistics | Ceftazidime-avibactam |
|--------------------------|------------|-----------------------|
| | | (N = xx) |
| DCCI Score | | |
| | n | xx |
| | Mean (SD) | xx x(xx xx) |
| | Median | xx x |
| | Min, Max | xx, xx |
| Comorbidities | | |
| Myocardial Infarction | | |
| Yes | n(%) | xx (xx x) |
| No | n(%) | xx(xxx) |
| Congestive Heart Failure | | |
| Yes | n(%) | xx (xx x) |
| No | n(%) | xx (xx x) |

 $Abbreviations: N = number \ of \ subjects \ in \ Ceftazidime-avibactam \ \ group; n = number \ of \ subjects \ in \ specified \ category$ 

DCCI= Deyo-Charlson Comorbidity Index

Note 1: Percentages are based on the number of subjects in the Ceftazidime-avibactam group.

Table 14.1.2.10 Indwelling Devices at the time of Infection Diagnosis – All Subejcts

| Indwelling Devices | Statistics | Ceftazidime-avibactam $(N = xx)$ |
|---|---|---|
| None | | |
| Intravenous peripheric catheter | n(%) | xx (xx x) |
| Intravenous central catheter | n(%) | xx (xx x) |
| Urinary catheter | n(%) | xx (xx x) |
| Any Drain | | |
| Site XXXXX | n(%) | xx(xxx) |
| Site XXXXX | n(%) | xx(xxx) |
| Other (Specify) | n(%) | xx (xx x) |

Abbreviations: N = number of subjects in Ceftazidime-avibactam group; n = number of subjects in specified category Note 1: Percentages are based on the number of subjects in the Ceftazidime-avibactam group.

Table 14.1.2.11 Disease Severity –All Subjects

| Disease Severity | Statistics | Ceftazidime-avibactam |
|--------------------------------|------------|-----------------------|
| | | (N = xx) |
| APACHE II Completed | | |
| Yes | n(%) | xx(xxx) |
| No | n(%) | xx(xxx) |
| APACHE Score | | |
| | n | XX |
| | Mean (SD) | xx x(xx xx) |
| | Median | xx x |
| | Min, Max | XX, XX |
| Another Disease Severity Score | | |
| Yes | n(%) | xx(xxx) |
| No | n(%) | xx(xxx) |
| Severity Score Used | | |
| XXXXXX | n(%) | xx (xx x) |
| XXXXXX | n(%) | xx (xx x) |
| Severity Score | | |
| | n | XX |
| | Mean (SD) | xx x(xx xx) |
| | Median | xx x |
| | Min, Max | xx, xx |

Abbreviations: N = number of subjects in Ceftazidime-avibactam group; n = number of subjects in specified category Note 1: Percentages are based on the number of subjects in the Ceftazidime-avibactam group.

Table 14.1.2.12 Source of Infection at Baseline – All Subjects

| Source of Infection | Statistics | Ceftazidime-<br>avibactam<br>(N = xx) |
|---|---|---|
| Hospital Acquired Infection (HAI) | n(%) | xx (xx x) |
| Healthcare Associated Infection (HCAI) | n(%) | xx (xx x) |
| CommunityAcquired Infection (CAI) | n(%) | xx(xxx) |

Abbreviations: N = number of subjects in Ceftazidime-avibactam group; n = Number of subjects in specified category.
Reference Listing xxxxx

Table 14.1.2.13 Indications and Reasons for Use of Ceftazidime-Avibactam- All Subjects

| Indications and Reasons | Statistics | Ceftazidime-<br>avibactam |
|---|---|---|
| | | (N = xx) |
| UTI | n(%) | xx (xx x) |
| Primary Diagnosis | | |
| xxxxxx | n(%) | xx (xx x) |
| xxxxxx | n(%) | xx (xx x) |
| Secondary Diagnosis | | |
| xxxxxx | n(%) | xx (xx x) |
| xxxxxx | n(%) | xx (xx x) |
| Symptoms | | |
| xxxxxx | n(%) | xx (xx x) |
| xxxxxx | n(%) | xx (xx x) |
| Positive dipstick for leukocyte esterase and/or nitrit | e | |
| Yes | n(%) | xx (xx x) |
| No | n(%) | xx (xx x) |
| Did the Patient have Secondary Bacteremia | | |
| Yes | n(%) | xx (xx x) |
| No | n(%) | xx (xx x) |
| Unknown | n(%) | xx (xx x) |
| IAI | n(%) | xx (xx x) |

Abbreviations: N = number of subjects in Ceftazidime-avibactam group; n = Number of subjects in specified category.

Table 14.2.1.1 Clinical Symptom Improvement –All Subjects

| Time point of Evaluation of ceftazidime-avibactam initiation | Clinical Symptom<br>Improvement | Statistics | Ceftazidime-avibactam $(N = xx)$ |
|---|---|---|---|
| 72 Hours (Day 3) | Symptom Assessment | | |
| | Symptom Improved | n (%) | xx(xxx) |
| | Symptom Worsened | n (%) | xx(xxx) |
| | Not Assesed | n (%) | xx (xx x) |
| Day 7 | Symptom Assessment | | |
| | Symptom Improved | n (%) | xx(xxx) |
| | Symptom Worsened | n (%) | xx(xxx) |
| | Not Assesed | n (%) | xx(xxx) |
| | Clinical Outcome | | |
| | Clinical Success | n (%) | xx (xx x) |
| | Clinical Failure | n (%) | xx (xx x) |
| | Clinical Indeterminate | n (%) | xx (xx x) |
| Day 14/EOT | | | |

Abbreviations: N = number of subjects in Ceftazidime-avibactam group; n = number of subjects in specified category; EOT=End of Treatment

Reference Listing xxxxxx

Programmer's Note 1: Consider Day 14 / End of Treatment, whichever is earlier.

Table 14.2.1.2 Microbiological Evaluation –All Subjects

| Time point of Evaluation of ceftazidime-avibactam initiation | Microbiological Evaluation | Statistics | Ceftazidime-avibactam $(N = xx)$ |
|---|---|---|---|
| Day 7 | Microbiological Success | n (%) | xx (xx.x) |
| | Microbiological Failure | n (%) | xx (xx.x) |
| | Microbiological Outcome | | |
| | Eradication | n (%) | xx (xx.x) |
| | Presumed Eradication | n (%) | xx (xx x) |
| | Verified Persistence | n (%) | xx (xx x) |
| Day 14/EOT | | | |

Abbreviations: N = number of subjects in Ceftazidime-avibactam group; n = number of subjects in specified category;

EOT=End of Treatment
Reference Listing xxxxxx
Table 14.2.2.3 Gram Negative Organisms Identified – All Subjects

| ram Negative Organisms Identified | Statistics | Ceftazidime-avibactam (N = $xx$ ) |
|---|---|---|
| Gram negative, Escherichi a Coli | n(%) | xx (xx x) |
| Gram negative, Klebsiella pneumonia | n(%) | xx (xx x) |
| Gram negative, Klebsiella spp | n(%) | xx (xx x) |
| Gram negative, Proteus mirabilis | n(%) | xx (xx x) |
| Gram negative, proteus spp | n(%) | xx (xx x) |

Abbreviations: N = number of subjects in Ceftazidime-avibactam group; n = Number of subjects in specified category.

Reference Listing xxxxxx

Programmer's Note 1: Continue the above table for all other gram negative identified bacteria.

Table 14.2.2.4 Susceptibility to Ceftazidime -Avibactam – All Subjects

| Susceptibility | Statistics | Ceftazidime-<br>avibactam (N =<br>xx) |
|-------------------------|------------|---------------------------------------|
| Susceptibility Organism | | |
| Xxxx | n (%) | xx(xxx) |
| Xxxx | n (%) | xx(xxx) |
| Xxxx | n (%) | xx(xxx) |
| | n (%) | xx (xx x) |
| Method used | | |
| E-test | n (%) | xx (xx x) |
| DISC | n (%) | xx (xx x) |
| If E-test, MIC value | n | XX |
| | Mean (SD) | xx xx (xx xxx) |
| | Median | XX XX |
| | Min, Max | xx x, xx x |
| If DISC, Zone Diameter | N | XX |
| | Mean (SD) | xx xx (xx xxx) |
| | Median | XX XX |
| | Min, Max | xx x, xx x |
| Susceptible | | |
| Yes | n (%) | xx (xx x) |
| No | n (%) | xx (xx x) |

Table 14.2.2.5 Length of Stay in Hospital/ICU – All Subjects

| Susceptibility | Statistics | Ceftazidime-<br>avibactam (N =<br>xx) |
|----------------|------------|---------------------------------------|
| Hospital LOS | n | XX |
| | Mean (SD) | xx xx (xx xxx) |
| | Median | xx xx |
| | Min, Max | xx x, xx x |
| ICU LOS | n | XX |
| | Mean (SD) | xx xx (xx xxx) |
| | Median | XX XX |
| | Min, Max | xx x, xx x |
| Susceptible | | |
| Yes | n (%) | xx (xx x) |
| No | n (%) | xx (xx x) |

Abbreviations: N = number of subjects in Ceftazidime-avibactam group; n = Number of subjects in specified category. LOS = Length of Stay

Hospital LOS is calculated as :1) the total number of consecutive days the patient was treated in the hospital from admission to discharge during their initial hospitalization; 2) the total number of days hospitalization between diagnosis of infection and discharge; 3) the total number of days the patient was treated in the hospital after ceftazidime-avibactam initiation up to hospital discharge, including the first day of treatment.

ICU LOS will be calculated as: 1) the total number of consecutive or non-consecutive days the patient was treated in the ICU during their initial hospitalization; and 2) the total number of days the patient was treated in the ICU after ceftazidime-avibactam initiation, including the first day of treatment.

Reference Listing xxxxxx

Table 14.3.1.1 Ceftazidime - Avibactam Exposure - All Subjects

| Ceftazidime - Avibactam Exposure | Statistics | Ceftazidime-avibactam |
|---|---|---|
| | | (N = xx) |
| Use of Ceftazidime-avibactam for >=48 hours reported in patient records? | | |
| Yes | n (%) | xx (xx x) |
| No | n (%) | xx (xx x) |
| Dose (mg) | N | XX |
| | Mean (SD) | xx x (xx xx) |
| | Median | xx x |
| | Min, Max | xx, xx |
| Frequency | | |
| BID | n(%) | xx (xx x) |
| OD | n(%) | xx (xx x) |
| Duration of Administration (hours) | N | xx |
| | Mean (SD) | xx x (xx xx) |
| | Median | xx x |
| | Min, Max | xx, xx |
| Category of Treatment | | |
| Empiric based on clinical judgement | n (%) | xx (xx x) |
| Empiric based on microbiology | n (%) | xx (xx x) |
| Reason for Discontinuation | | |
| Adverse Events | n (%) | xx (xx x) |
| Perceived Clinical Failure | n (%) | xx (xx x) |
| Total Duration of therapy (days) | N | XX |
| | Mean (SD) | xx x (xx xx) |

Program Name: Txx.sas Produced: DDMMMYYYY

Reference Listing xxxxxx

| Median | xx x |
|---|---|
| Min, Max | xx, xx |
| Abbreviations: $N = \text{number of subjects in Ceftazidime-avibactam group}$ ; $n = Nu$ | imber of subjects in specified category. |

Table 14.3.2.1 Summary of Subjects with AEs -All Subjects

| | Statistics $(N = xx)$ | Ceftazidime-avibactam |
|---|---|---|
| | | (N = xx) |
| Subjects with Adverse Events | n (%) | xx ( xx.x) |
| Subjects with Serious AEs | n (%) | xx (xx.x) |
| AE related to | | |
| Ceftazidime-avibactam | n (%) | xx ( xx.x) |
| Concomitant medication | n (%) | xx ( xx.x) |
| Other pfizer drug | n (%) | xx (xx.x) |
| Serious AE related to | | |
| Ceftazidime-avibactam | n (%) | xx ( xx.x) |
| Concomitant medication | n (%) | xx ( xx.x) |
| Other pfizer drug | n (%) | xx (xx.x) |
| Outcome of the AEs | | |
| Recovered/Resolved | n (%) | xx ( xx.x) |
| Recovered/Resolved with sequelae | n (%) | xx ( xx.x) |
| Recovering/Resolving | n (%) | xx ( xx.x) |
| Not Recovered/Not Resolved | n (%) | xx ( xx.x) |
| Fatal | n (%) | xx (xx.x) |
| Action Taken withdrawn | | |
| Dose Reduced | n (%) | xx (xx.x) |
| Dose Increased | n (%) | xx (xx.x) |
| Dose not changed | n (%) | xx (xx.x) |
| Unknown | n (%) | xx ( xx.x) |

Abbreviations: N = number of subjects in Ceftazidime-avibactam group; n = number of subjects in specified category
Note 1: Percentages are based on number of subjects in respective treatment groups
Reference Listing xxxxxx

Program Name: Txx.sas Produced: DDMMMYYYY

Table 14.3.2.2 Summary of Subjects With AE's by Soc And PT- All Subjects

| System Organ Class | Statistics | Ceftazidime-avibactam |
|---------------------------------|------------|-----------------------|
| Preferred Term | | (N = xx) |
| Subjects having at least one AE | n (%) | xx ( xx.x) |
| System Organ Class 1 | n (%) | xx ( xx.x) |
| Preferred Term 1 | n (%) | xx ( xx.x) |
| Preferred Term 2 | n (%) | xx ( xx.x) |
| Preferred Term 3 | n (%) | xx ( xx.x) |
| System Organ Class 2 | n (%) | xx ( xx.x) |
| Preferred Term 1 | n (%) | xx (xx.x) |
| Preferred Term 2 | n (%) | xx ( xx.x) |

Abbreviations: N = number of subjects in Ceftazidime-avibactam group; n = number of subjects in specified category

Note 1: System organ class and preferred terms are coded using the standards of MedDRA xxxx

Note 2: Percentages are based on number of subjects in treatment group

Reference Listing xxxxxx

Programmer's Note 1: System organ classes and Preferred Terms are sorted in descending order of frequency in Ceftazidime-avibactam.

Programmer's Note 2: The table will continue for all other SOC and PT.

Programmer's Note 3: Similar tables will be generated as follows:

Table 14.3.2.3 Summary of Subjects with Serious AEs by SOC and PT – All Subjects

Table 14.3.2.4 Summary of Subjects with Study Drug Related AEs by SOC and PT – All Subjects

Table 14.3.2.5 Summary of Subjects with other Pfizer Drug Related AEs by SOC and PT – All Subjects

Table 14.3.2.6 Summary of Subjects with AEs leading to death by SOC and PT – All Subjects

Table 14.3.2.7 Summary of Subjects with AEs leading to permanent discontinuation of study drug by SOC and PT -All Subjects

Table 14.3.3.1 Recurrence of Infection – All Subjects

| Symptoms | Statistics | Ceftazidime-<br>avibactam (N =<br>xx) |
|---|---|---|
| Recurrence of infection | | |
| Yes | n (%) | xx (xx x) |
| No | n (%) | xx (xx x) |
| If yes, site of infection/micro-organism | ı | |
| Same | n (%) | xx (xx x) |
| Different | n (%) | xx (xx x) |
| If Different, New site of infection | | |
| Xxxx | n (%) | xx(xxx) |
| Xxxx | n (%) | xx(xxx) |
| Xxxx | n (%) | xx(xxx) |
| If Different, Micro-organism | | |
| Xxxx | n (%) | xx (xx x) |
| Xxxx | n (%) | xx (xx x) |
| Xxxx | n (%) | xx (xx x) |

Program Name: Txx.sas Produced: DDMMMYYYY

Table 14.3.4.1 Microbiology Results- All Subjects

| Timing of sample collection | Pathogens identified | Statistics | Ceftazidime-avibactan<br>(N=xx) |
|---|---|---|---|
| Before initial antibiotic therapy | No. of Bacterial Pathogens Identified | | |
| Before initial antibiotic therapy | No. of Bacterial Fathogens Identified | n<br>Maan (SD) | XX |
| | | Mean (SD) | xx xx (xx xxx) |
| | | Median | XX XX |
| | | Min, Max | XX X, XX X |
| | Bacterial Pathogen Identified | | |
| | Gram negative, Escherichi a Coli | n(%) | xx (xx x) |
| | Gram negative, Klebsiella pneumonia | n(%) | xx (xx x) |
| | Gram negative, Klebsiella spp | n(%) | xx (xx x) |
| | Fungal Pathogen, if identified | | |
| | XXXXXXX | n(%) | xx (xx x) |
| | XXXXXXX | n(%) | xx (xx x) |
| After initial antibiotic therapy but before | | | |
| ceftazidimeavibactam therapy | | | |

Table 14.3.5.1 Pathogen Susceptibility – All Subjects

| Pathogen<br>Sensitivity | Statistics | Ceftazidime-<br>avibactam<br>(N = xx) |
|---|---|---|
| Communities Education Colli | (0.1) | |
| Gram negative, Esherichia Coli | n(%) | xx (xx x) |
| Susceptible | n(%) | xx(xxx) |
| Intermediate | n(%) | xx(xx) |
| Resistant | n(%) | xx(xxx) |
| xxxxxxxxx | n(%) | xx ( xx x) |
| | n(%) | xx(xx) |
| | n(%) | xx(xxx) |

-----

Table 14.3.6.1 In-Hospital Mortality – All Subjects

| | Statistics | Ceftazidime-avibactam $(N = xx)$ |
|-----------------------|------------|----------------------------------|
| In-Hospital Mortality | | |
| Yes | n (%) | xx ( xx.x) |

Abbreviations: N = number of subjects in Ceftazidime-avibactam group; n = number of subjects in specified category

Note 1: Percentages are based on number of subjects in treatment group.

Reference listing xxxxxxx

Program Name: LXX.sas Produced: DDMMMYYYY

### **Appendix 10.2 Mock Shells for Listings**

General Notes for programmers:

1. For more details regarding listings please refer to SAP write-up, protocol, CRF and metadata.

2. If there are no counts in any of the listings then display the line "No Patient Meets the Reporting Criteria" in the body of listing.

3. The title on each listing is as follows

Protocol Number: X9001260 Status=SHELLS Page X of Y

Program Name: LXX.sas Produced: DDMMMYYYY

Whereas Status of the report should be Shells (at Draft stage) and change to Final (for Final output)

4. Report should be produced with "Times New Roman" as text font and height of the text should be 9.

5. Report should have Left, Right, Top and Bottom Margins to 1.

6. Footnote text mentioned in Mock Shell starts with "Programmer's Note": is only a note for Programmer and is not a part of Report.

- 7. Footnote text mentioned in Mock Shell starts with "Note" will be presented as footnote during generation of listings .
- 8. In the listing wherever appropriate please replace the /<Event Nr.> with the actual value.

Page X of Y

# Table of Contents

| Listing 16.2.1.1 Site Characteristics— All subjects data | 3 |
|---|---|
| Listing 16.2.1.2 Local Gram-negative Resistance Patterns – All Subjects Data | 4 |
| Listing 16.2.1.3 Demographic Characteristics – Safety Population | 5 |
| Listing 16.2.2.1 Renal Status of Patient – Safety Population | 6 |
| Listing 16.2.2.2 Comorbidities (Deyo-Charlson Comorbidity Index) – All Subjects | 7 |
| Listing 16.2.2.3 Disease Severity – All Subjects | 8 |
| Listing 16.2.2.4 Additional Risk Factor -All Subjects | 9 |
| Listing 16.2.3.1 Index Hospitalization -All Subjects | 10 |
| Listing 16.2.3.2 Length of Hospital Stay – Safety Population | 11 |
| Listing 16.2.3.3 Current Admission to ICU – All Subjects | 12 |
| Listing 16.2.3.4 Prior Recent Hospitalization -Safety Population | 13 |
| Listing 16.2.3.5 Recent Healthcare Procedures -Safety Population | 14 |
| Listing 16.2.3.6 Healthcare Utilization – Safety Population | 15 |
| Listing 16.2.4.1 Indication – All Subjects | 16 |
| Listing 16.2.5.1 Ceftazidime-Avibactam Exposure – All Subjects | 17 |
| Listing 16.2.5.2 History of Prior Antibiotic Exposure – All Subject Data | 18 |
| Listing 16.2.5.3 Concomitant Antibiotic Therapy – All Subject Data | 19 |
| Listing 16.2.5.4 Antibiotic Therapy: Prior lines of Treatment – All Subjects | 19 |
| Listing 16.2.5.5 Antibiotic Treatment After Ceftazidime-Avibactam All Subjects | 19 |
| Listing 16.2.6.1 Clinical Symptoms Improvement– All Subjects | 20 |
| Listing 16.2.6.2 Microbiological Evaluation - Safety Population | 21 |
| Listing 16.2.6.3 Recurrence of Infection – Safety Population | 22 |
| Listing 16.2.6.4 Susceptibility to Ceftazidime-Avibactam – All Subjects | 23 |
| Listing 16.2.7.1 Microbiology– All Subjects | 24 |
| Listing 16.2.7.2 Pathogen Susceptibility – Safety Population | 25 |
| Listing 16.2.8.1 In-Hospital Mortality – Safety Population | 26 |
| Listing 16.2.9.1 Adverse Events – Safety Population | 27 |

Listing 16.2.1.1 Site Characteristics—All subjects data

| Unique Subject ID | Physician Specialty | | Hos | Hospital Information | |
|---|---|---|---|---|---|
| | Medical specialty of<br>the treating<br>physician | Care Level | Hospital Type | Total number of beds | Total number of ICU beds |
| xxxx-xxxx | XXXX | Secondary | Teaching | XXX | XX |
| хххх-хххх-хххх | xxxx | Tertiary | Teaching | xxx | XX |

Programmer's Note 1: This listing will continue for all site and subjects will be sorted in ascending order by unique Subject ID.

Program Name: LXX.sas Produced: DDMMMYYYY

Listing 16.2.1.2 Local Gram-negative Resistance Patterns – All Subjects Data

| Unique Subject ID | Is the percentage of gram-negative isolates that exhibit resistance to 3rd generation known for: | Rate available between 01<br>June 2019 and 01 April<br>2020, rate (%)/ Rate<br>available over a different<br>time period, rate (%) | Rate(%) | Time period start date/time period end date |
|---|---|---|---|---|
| xxxx-xxxx | Cephalosporins | Rate available between 01<br>June 2019 and 01 April<br>2020, rate (% | xx | DDMMMYYYY/DDMMMYYYY |
| xxxx-xxxx | Carbapenem | Rate available between 01<br>June 2019 and 01 April<br>2020, rate (% | xx | DDMMMYYYY/DDMMMYYYY |

Programmer's Note 1: This listing will continue for all subjects and antibiotics and will be sorted in ascending order by unique Subject ID.

Program Name: LXX.sas Produced: DDMMMYYYY

**Listing 16.2.1.3 Demographic Characteristics – All Subjects Data** 

| Unique Subject ID | Year of Birth | Gender | Age (Years) | Height(cm) | Weight(kg) | Current employment status |
|---|---|---|---|---|---|---|
| xxxx-xxxx | YYYY | Male | XX | Xxx | xx | Full Time |
| xxxx-xxxx | YYYY | Female | xx | XXX | xx | Part time |

Program Name: LXX.sas Produced: DDMMMYYYY

**Listing 16.2.2.1 Renal Status of Patient – All Subjects Data** 

| Unique Subject ID | Serum Creatinine (mg/dl) | CRCL (ml/min) | Severity of renal dysfunction |
|---|---|---|---|
| xxxx-xxxx | xx xx | xx xx | Mild |
| xxxx-xxxx | xx xx | xx xx | Severe |

Note 1: Subjects with renal dysfunction have been listed.

Programmer's Note 1: The above listing will be continued for all the other subjects order by Unique Subject ID.

Program Name: LXX.sas Produced: DDMMMYYYY

Listing 16.2.2.2 Comorbidities (Deyo-Charlson Comorbidity Index) – All Subjects Data

| Unique<br>Subject ID | Comorbidity | Deyo-<br>Charlson<br>Comorbidity<br>Index | Deyo-<br>Charlson<br>Weight | Diagnosis | Diagnosis date | Chemotherapy<br>received in last<br>three months | Location of<br>other<br>transplant | Glasgow<br>coma score |
|---|---|---|---|---|---|---|---|---|
| xxxx-xxxx-<br>xxxx | Myocardial<br>Infarction | 2 | 1 | - | | | | |
| | Malignancy | 2 | 6 | Solid tumor | DDMMMYYYY | Yes | | |

Note 1: Subjects with at least one comorbidity conditions have been listed.

Programmer's Note 1: The above listing will be continued for all other comorbidity and subjects will be sorted in ascending order by Unique Subject ID.

Program Name: LXX.sas Produced: DDMMMYYYY

**Listing 16.2.2.3 Disease Severity – All Subjects Data** 

| Unique Subject ID | Was APACHE II completed? | Score | Was another disease severity score completed? | If Yes, name of severity score | Score |
|---|---|---|---|---|---|
| | 37 | | | | |
| XXXX-XXXX-XXXX | Yes | Xx | Yes | XXXX | XX |
| XXXX-XXXX-XXXX | Yes | XX | No | - | |
| Note 1: Subjects with a | at least one severity score | have been listed. | | | |

Program Name: LXX.sas Produced: DDMMMYYYY

Listing 16.2.2.4 Additional Risk Factor - All Subjects Data

| Unique<br>Subject ID | Has patient<br>travelled to any<br>foreign country<br>in the last 3<br>months? | If Yes,<br>provide<br>country | Start Date/<br>Return Date | Was subject hospitalized during travel? | Is the patient pregnant?? | No. of weeks<br>of gestation<br>since last<br>menstrual<br>period | Does patient drink alcohol ? | No. of<br>drink per<br>week | Tobacc<br>o Use | Cigarettes<br>per day/No.<br>of years<br>smoking | No. of<br>Years<br>Smoking |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXX-XXXX-<br>XXX | Yes | xxxxxx | DDMMMYYY<br>Y/<br>DDMMMYYY<br>Y | No | NA | - | No | - | Current<br>Smoker | 5 | 10 |
| XXXX-XXXX-<br>XXX | No | | | | Yes | xx | No | - | Never<br>Smoked | | |

Programmer's Note 1: The above listing will be continued for all other subjects ascending order by Unique Subject ID and visit.

Program Name: LXX.sas Produced: DDMMMYYYY

Listing 16.2.3.1 Index Hospitalization - All Subjects Data

| Unique<br>Subject ID | Date of index<br>hospitalization<br>admission | Mode of admission | Source of admission | Ward<br>admitted<br>for initial<br>hospitalizat<br>ion | Diagnosis at admission | Was the patient discharged by the end of the study period? | Date of<br>hospital<br>discharge | Ward<br>admitted | Ward<br>admission<br>date | Ward<br>discharge/<br>transfer date |
|---|---|---|---|---|---|---|---|---|---|---|
| xxxx-xxxx-<br>xxx | DDMMMYYYY | Emergency | Outpatient | Surgical | xxxxx | Yes | DDMMMY<br>YYY | I-Ward | DDMMMY<br>YYY | DDMMMYY<br>YY |
| XXXX-XXXX-<br>XXX | DDMMMYYYY | Scheduled | Long term care facility | Medical | XXXXX | No | DDMMMY<br>YYY | | | |

Programmer's Note 1: The above listing will be continued for all other subjects ascending order by Unique Subject ID

Program Name: LXX.sas Produced: DDMMMYYYY

Listing 16.2.3.2 Length of Hospital Stay – All Subjects Data

| Unique Subject ID | Date(s) of<br>hospital<br>admission | Date(s) of<br>hospital<br>discharge | Patient admitted in ICU? | IF Yes, Date of ICU admission | IF Yes, Date of<br>ICU discharge | If yes, Diagnosis at admission |
|---|---|---|---|---|---|---|
| xxxx-xxxx-xxx | DDMMMYYYY | DDMMMYYYY | Yes | DDMMMYY<br>YY | DDMMMYYYY | xxxxxxxx |
| xxxx-xxxx | DDMMMYYYY | - | No | | - | |
| Programmer's Note 1: | The above listing will | be continued for all | other subjects and sorted i | n ascending order | by Unique Subject ID. | |

Program Name: LXX.sas Produced: DDMMMYYYY

Listing 16.2.3.3 Current Admission to ICU – All Subjects Data

| Unique Subject ID | Reason for admission to ICU | Date of ICU admission | Date of ICU discharge | Date of Discharge from hospital |
|---|---|---|---|---|
| xxxx-xxxx | xxxxxx | DDMMMYYYY | DDMMMYYYY | DDMMMYYYY |
| xxxx-xxxx-xxxx | xxxxxxx | DDMMMYYY | DDMMMYYYY | |

Program Name: LXX.sas Produced: DDMMMYYYY

#### Listing 16.2.3.4 Prior Recent Hospitalization - All Subjects Data

| Unique Subject ID | Date of admission | Date of discharge | Reason for hospitalization/ Primary diagnosis at discharge |
|---|---|---|---|
| xxxx-xxxx | DDMMMYYYY | DDMMMYYYY | xxxxx |
| xxxx-xxxx | DDMMMYYYY | DDMMMYYYY | Xxxxx |

Note: Only subjects with recent hospitalization within 90 days prior to date of admission for the current hospitalization has been listed.

Programmer's Note 1: This listing will continue for all subjects and will be sorted in ascending order by unique Subject ID.

Protocol Number: X9001260 Page X of Y Status=SHELLS

Program Name: LXX.sas Produced: DDMMMYYYY

Listing 16.2.3.5 Recent Healthcare Procedures - All Subjects Data

| Unique Subject ID | Date of<br>healthcare procedure | Type of healthcare procedure |
|---|---|---|
| xxxx-xxxx | DDMMMYYYY | xxxxx |
| xxxx-xxxx | DDMMMYYYY | xxxxx |

Note: Only subjects with prior healthcare procedures within 30 days prior to ceftazidime-avibactam initiation have been listed.

Programmer's Note 1: This listing will continue for all subjects and will be sorted in ascending order by unique Subject ID.

Listing 16.2.3.6 Healthcare Utilization – All Subjects Data

| Unique Subject ID | Healthcare resource | Start date | Stop date | Details |
|---|---|---|---|---|
| xxxx-xxxx-xxx | Mechanical ventilation | DDMMMYYYY | DDMMMYYYY | xxxxxxx |
| xxxx-xxxx-xxx | Hemodialysis | DDMMMYYYY | DDMMMYYYY | xxxxxxx |

Note 1: Subjects with any use of healthcare resources during the initial hospitalization

Programmer's Note 1: The above listing will be continued for all other subjects and sorted in ascending order by Unique Subject ID.

Program Name: LXX.sas Produced: DDMMMYYYY

**Listing 16.2.4.1 Indication – All Subjects Data** 

| Unique<br>Subject<br>ID | Source of<br>Infection | Indication<br>for<br>ceftazidime-<br>avibactam | Primary<br>Diagnosis of<br>Indication | Secondary<br>Diagnosis<br>of<br>Indication | Symptoms | Date of<br>sampling | Positive dipstick for leukocyte esterase and/or nitrite | Date of diagnosis | Did the patient have a secondary bacteremia? | Explain<br>other; initial<br>site of<br>infection<br>(organ) |
|---|---|---|---|---|---|---|---|---|---|---|
| xxxx-<br>xxxx-xxxx | Hospital<br>Acquired<br>Infection (HAI) | UTI | Obstruction | Renal<br>failure | Fever | DDMMMYYYY | Yes | DDMMMYYYY | Yes | |
| | , , | IAI | Liver abscess | Pancreatic abscess | Hypothermi<br>a | | | DDMMMYYYY | | |
| | | NP | Hospital<br>Acquired<br>Pneumonia | | Fever | | | DDMMMYYYY | No | |
| | | Other | | | | | | | Yes | Appendix |
| XXXX-<br>XXXX-XXXX | | | | | | DDMMMYYY | | | | |

Note 1: Subjects with indication for ceftazidime-avibactam have been listed.

Program Name: LXX.sas Produced: DDMMMYYYY

## Listing 16.2.5.1 Ceftazidime-Avibactam Exposure – All Subjects Data

| Unique<br>Subject ID | Use of Ceftazidime-avibac tam for >=48 hours reported in patient records? | Start date/Stop<br>Date | Dose(mg) | Frequency | Route | Duration of<br>administratio<br>n (hours) | Category of treatment | Reason for discontinue | Total duration of therapy |
|---|---|---|---|---|---|---|---|---|---|
| xx-xxxx-xxxx | Yes | DDMMMYYYY/<br>DDMMMYYYY | XX | BD | IV | XX | empiric based on microbiology | Adverse<br>Event | xx |
| xx-xxxx-xxxx | Yes | DDMMMYYYY/<br>DDMMMYYYY | xx | OD | IV | XX | empiric based on<br>genotyping | Cure | XX |

-----

Programmer's Note: This listing will continue for all subjects and will be sorted in ascending order by unique Subject ID.

Listing 16.2.5.2 History of Prior Antibiotic Exposure – All Subject Data

| Unique<br>Subject ID | Antibiotic(s) used | Start date/Stop<br>Date | Dose(mg) | Frequency | Route | Reason for<br>Treatment<br>specify (if<br>available) |
|---|---|---|---|---|---|---|
| xx-xxxx-xxxx | xxxxxxx | DDMMMYYYY/ | xx | BID | IV | XX |
| | xxxxxxx | DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY | XX | OD | IV | XX |
| | xxxxxxxx | DDMMMYYYY/<br>DDMMMYYYY | XX | OD | IV | xx |
| xx-xxxx-xxxx | | | | | | |

Note 1: Subject with any antibiotic(s) used within 90 days prior to date of admission for the current hospitalization have been listed Programmer's Note: This listing will continue for all subjects and will be sorted in ascending order by unique subject Id.

Protocol Number: X9001260 Page X of Y Status=SHELLS

Program Name: LXX.sas Produced: DDMMMYYYY

Listing 16.2.5.3 Concomitant Antibiotic Therapy – All Subject Data

| Unique<br>Subject ID | Antibiotic(s) used | Start date/Stop<br>Date | Dose(mg) | Frequency | Route | Duration of administration (hours) | Category of treatment | Reason for discontinuati on |
|---|---|---|---|---|---|---|---|---|
| xx-xxxx-xxxx | Amikacin | DDMMMYYYY/<br>DDMMMYYYY | xx | BID | Oral | xx | empiric based on<br>microbiology | Adverse Event |
| | Amoxicillin | DDMMMYYYY/<br>DDMMMYYYY | XX | OD | Oral | XX | empiric based on genotyping | Cure |
| | Amoxicillin-<br>clavulanate | DDMMMYYYY/<br>DDMMMYYYY | XX | OD | Oral | XX | empiric based on genotyping | Adverse Event |
| xx-xxxx | clavulanate | | XX | OD | Oral | XX | - | |

Note 1: Subject with any antibiotic(s) used concurrently with ceftazidime-avibactam have been listed

Programmer's Note: This listing will continue for all subjects and will be sorted in ascending order by unique subject Id.

Programmer's Note 2: This similar listing will be generated as follows:

**Listing 16.2.5.4 Antibiotic Therapy: Prior lines of Treatment – All Subjects** Listing 16.2.5.5 Antibiotic Treatment After Ceftazidime-Avibactam All Subjects

Listing 16.2.6.1 Clinical Symptoms Improvement– All Subjects

| Unique Subject ID | Time point of evaluation of ceftazidime-avibactam initiation | Date of<br>evaluation | Symptom improved<br>or worsened (as reported<br>by physician) | Clinical outcomes |
|---|---|---|---|---|
| xx-xxxx-xxxx | Day 3 | DDMMMYYYY | Symptom improved | - |
| | Day 7 Day 14/ EOT Other | DDMMMYYYY | Symptom improved | Clinical Success |
| | | | nd all available time points will b | |

Programmer's Note: This listing will continue for all subjects and all available time points will be sorted in ascending order by unique subject ID

Program Name: LXX.sas Produced: DDMMMYYYY

**Listing 16.2.6.2 Microbiological Evaluation - All Subjects Data** 

| Unique Subject ID | Time point of evaluation of ceftazidime-avibactam initiation | Date of<br>evaluation | Microbiological<br>evolution | Microbiological<br>outcomes |
|---|---|---|---|---|
| xx-xxxx-xxxx | Day 7 | DDMMMYYYY | Microbiological success | Eradication |
| | Day 14/ EOT<br>Other | DDMMMYYYY | Microbiological success | Verified Persistence |

Program Name: LXX.sas Produced: DDMMMYYYY

**Listing 16.2.6.3 Recurrence of Infection – All Subjects Data** 

| Unique Subject ID | Was the site of infection/micro-<br>organism same or different? | If same, Micro<br>organisms | If different, New site of infection/ micro organisms |
|---|---|---|---|
| xxxx-xxxx | Same | xxxxxxxx | |
| xxxx-xxxx | Different | - | xxxxx/xxxxxx |
| Note 1:Subjects with syr 30 days have been listed | mptoms and signs of a new infection after | completion of treatment | t with Ceftazidime avibactam till |

Programmer's Note 1: The above listing will be continued for all other subjects and sorted in ascending order by Unique Subject ID.

Listing 16.2.6.4 Susceptibility to Ceftazidime-Avibactam – All Subjects

| Unique Subject ID | Date of susceptibility testing | Organism | Method used | MIC value/ Zone<br>diameter | Susceptible |
|---|---|---|---|---|---|
| xxxx-xxxx | DDMMMYYYY<br>DDMMMYYYY | Xxxxx<br>Xxxxx | E-test<br>DISC | Xxx<br>xxxx | Yes<br>No |

Note 1: Subjects with susceptibility testing done have been listed.

Programmer's Note 1: The above listing will be continued for all the other subjects, visits and sorted in ascending order by Unique Subject ID and Visit

Program Name: LXX.sas Produced: DDMMMYYYY

### Listing 16.2.7.1 Microbiology- All Subjects

| Unique Subject<br>ID | Timing of sample collection | Date of identification | Number of<br>bacterial<br>pathogens<br>identified | Specify<br>fungal<br>Pathoge<br>n if<br>identifie<br>d | Type of<br>specime<br>n | Bacterial<br>pathogens<br>identified | Name of the pathogen/Site | Do the bacteria present any beta lactamase? | Genotyping<br>Done/How<br>many were<br>identified? | Name and<br>Class of Beta<br>Lactamase |
|---|---|---|---|---|---|---|---|---|---|---|
| xxxx-xxxx | Before initial antibiotic therapy | DDMMMYYYY | Unknown | xxxxxx | Blood | Gram negative,<br>Escherichia<br>Coli | xxxx/Urine | Yes | Yes/2 | extended<br>spectrum B<br>lactamase |
| | After initiation or during ceftazidime-avibactam therapy | DDMMMYYYY | XXX | | Blood | Gram negative,<br>Escherichia<br>Coli | xxxx/Blood | Unknown | No | |

-----

Note 1: Subjects with microbiology sample taken have been listed.

Programmer's Note 1: The above listing will be continued for all the other subjects, visits and sorted in ascending order by Unique Subject ID and Visit

Listing 16.2.7.2 Pathogen Susceptibility – All Subjects Data

| Unique Subject ID | Pathogen | Name of the Pathogen | Date of Pathogen | Sensitivity | Drug |
|---|---|---|---|---|---|
| xxxx-xxxx-xxx | Gram negative,<br>Esherichia Coli | xxxxxxxxx | DDMMMYYYY | S -3 | Xxxxx<br>Xxxxxx<br>Xxxxxx<br>Xxxxxxx |
| | Gram negative,<br>Proteus spp | xxxxxxxxx | DDMMMYYYY | R -2 | Xxxxxx<br>Xxxxxx<br>Xxxxxx |

Note 1: Subjects with any of the pathogens identified susceptible to antibiotics have been listed.

Programmer's Note 1: The above listing will be continued for all the other subjects, visits and sorted in ascending order by Unique Subject ID and Visit

Program Name: LXX.sas Produced: DDMMMYYYY

## Listing 16.2.8.1 In-Hospital Mortality – All Subjects Data

| Unique Subject ID | Date of death | Cause of death | |
|---|---|---|---|
| | 2210000000 | | |
| XXXX-XXXX-XXX | DDMMMYYYY | XXXXXX | |
| xxxx-xxxx-xxx | DDMMMYYYY | xxxxxxx | |
| Note 1: Only subjects died during h | ospitalization have been listed | | |
| Programmer's Note 1: The above li Subject ID. | sting will be continued for all other subje | ects and sorted in ascending order by U | Unique |

Program Name: LXX.sas Produced: DDMMMYYYY

#### Listing 16.2.9.1 Adverse Events – All Subjects Data

| Unique Subject<br>ID | AE Term | SOC/PT | Start Date/ Stop<br>Date/ Ongoing | Relationship | AE Serious<br>(Yes/No) | Criteria for seriousness | Outcome | Action<br>taken for AE |
|---|---|---|---|---|---|---|---|---|
| xxxx-xxxx | xxxxx | xxxxxx/xxxxxx | DDMMMYYYY/<br>DDMMMYYYY | Ceftazidime-<br>avibactam | No | Life<br>Threatening | Recovering /<br>Resolving | Dose not changed |
| | xxxxxx | xxxxx/xxxxxx | DDMMMYYYY/<br>DDMMMYYYY | Concomitant drug | Yes | Fatal | Fatal | Unknown |

Note 1: AE = Adverse Event, SOC = System Organ Class, PT = Preferred Term

Note 2: SOC and PT are coded using latest version of MedDRA dictionary.

Note 3: Only subjects with at least one adverse event are listed.

Programmer's Note 1: The listing will continue for all other subjects with AEs and sorted in ascending order by Unique Subject ID and Visit.